CLINICAL TRIAL: NCT02180789
Title: An Open-label, Prospective Interventional Study of the Tolerability and Efficacy of Oral Harnalidge® OCAS® (Tamsulosin) 0.4 mg in Patients Who Are Unsatisfied With the Treatment of Tamsulosin 0.2 mg
Brief Title: A Study to Evaluate the Tolerability and Efficacy of Tamsulosin 0.4mg OCAS Formulation in Patients Who Are Unsatisfied With the Treatment of Tamsulosin 0.2mg Conventional Formulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAURO-1201-TW
Record Dates: First submitted 2014-06-25; First posted 2014-07-03 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Lower Urinary Tract Symptoms (LUTS) Associated With Benign Prostatic Hyperplasia (BPH)
Keywords: tamsulosin,; benign prostatic hyperplasia,; α1-adrenoceptor antagonists
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Harnalidge® OCAS® (Experimental)
  Interventions: Drug: Tamsulosin OCAS

INTERVENTIONS:
Drug: Tamsulosin OCAS — oral
  Other Names: Harnalidge® OCAS®

SUMMARY:
This is an open-label, single-arm, prospective interventional study to assess the tolerability and efficacy of Harnalidge® OCAS® 0.4 mg in Taiwan patients who are unsatisfied with tamsulosin 0.2 mg for the treatment of lower urinary tract symptoms (LUTS) associated with benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
After obtaining informed consent, subjects who meet the inclusion criteria and not violating the exclusion criteria will be enrolled to receive Harnalidge® OCAS® 0.4 mg for treatment. The interventional period for the study is three months after the first date of enrollment or until the patients are discontinued the treatment of Harnalidge® OCAS®. All subjects will be instructed to contact the site if a patient's partner becomes pregnant during or within 90 days from the discontinuation of dosing, the investigator should report the information to the sponsor as if it is an SAE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as LUTS associated with BPH
* Currently taking oral tamsulosin 0.2 mg for at least 4 weeks
* Unsatisfied with the treatment of tamsulosin 0.2 mg The definition of 'unsatisfaction' is based on patient's satisfaction. Investigator will ask patient one question "Are you satisfied with your current treatment?" prior to study enrollment
* IPSS-QOL score ≧3 points at baseline

Exclusion Criteria:

* Subjects who underwent prostatectomy during the period of one year prior to this study
* Subjects with neurogenic bladder dysfunction, bladder neck sclerosis, urethral stricture, prostatic cancer, cystolithiasis, severe vesical diverticulum, urinary tract infection
* Subjects with any other complication which may cause voiding dysfunction
* Subjects with severe hepatic dysfunction, severe renal dysfunction, severe cardiovascular disorders, orthostatic hypotension, or senile dementia
* Subjects clinically significant condition, which in the opinion of the investigator makes the patients unsuitable for the trial
* Subjects who are currently participating in any other investigational drug study or who have participated in a study of an investigational drug within 3 months prior to this study

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in total scores of International Prostate Symptom Score (IPSS) | baseline, 4-week, 8-week, 12 week

SECONDARY OUTCOMES:
Changes from baseline in IPSS subscore | baseline, 4-week, 8-week, 12 week
  IPSS subscores include storage subscores, voiding subscores and nocturia
Changes from baseline in total scores of Quality of life (QOL) index (IPSS-QOL) | baseline, 4-week, 8-week, 12 week
Changes from baseline in Uroflowmetry parameters | baseline, 4-week, 8-week, 12 week
  Uroflowmetry parameters include Qmax, Qave, and voided volume
Changes from baseline in Visual Analogue Scale (VAS) | baseline, 4-week, 8-week, 12 week
  VAS is a vertical mark on a 10-cm line that ran from 'Not at all' to 'Yes, completely'. Patient marks on the line the point that they feel represents their perception of treatment satisfaction; 'Not at all' = 0 to 'Yes, completely' =10
Safety assessed by the adverse events, physical examination, vital signs and post void residual volume | Up to 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Linkou District, Taiwan

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=HAURO-1201-TW